CLINICAL TRIAL: NCT07025889
Title: IBI343 Combined With Sintilimab Plus Chemotherapy in Previously Untreated, Claudin (CLDN) 18.2-positive, HER2-negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (Dragon15)
Brief Title: IBI343 Combined With Sintilimab Plus Chemotherapy in Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dragon15
Record Dates: First submitted 2025-06-05; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; IBI 343; Sintilimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): IBI343 Combined with Sintilimab Plus SOX
  Interventions: Drug: IBI343; Drug: Sintilimab; Drug: Oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: IBI343 — Subjects in the phase 1b stage will receive IBI343 3/4.5/6mg/kg intravenous infusion (IV) D1 Q3W in 3-week cycles.
  Subjects in the phase 2 stage will receive IBI343 RP2D intravenous IV D1 Q3W in 3-week cycles.
Drug: Sintilimab — Subjects will receive sintilimab 200mg IV D1 Q3W in 3-week cycles.
Drug: Oxaliplatin — Subjects will receive oxaliplatin 130mg/m2 IV D1 Q3W in 3-week cycles.
Drug: S-1 — Subjects will receive S-1 40-60mg BID PO D1-14 Q3W in 3-week cycles.

SUMMARY:
This is a Single-arm, Open-label, Phase 1b/2 Study of IBI343 Combined with Sintilimab Plus Chemotherapy in Previously Untreated, Claudin (CLDN) 18.2-positive, HER2-negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma

DETAILED DESCRIPTION:
This trial is a phase Ib/II study to evaluate the safety, tolerability and efficacy of IBI343 in combination with sintilimab and chemotherapy in patients with advanced gastric or gastroesophageal junction (G/GEJ) adenocarcinoma. In dose-escalation stage, patients with CLDN 18.2-positive, HER2-negative were treated with IBI 343, sintilimab, and chemotherapy (oxaliplatin, S-1) as first-line therapy, which followed a 3+3 design. The dose expansion stage aimed to further investigate the safety and preliminary efficacy of recommended phase II dose (RP2D), including Cohort 1 and Cohort 2. In Cohort 1, 25 patients with CLDN18.2-positive, HER2-negative advanced G/GEJ adenocarcinoma will be enrolled. In Cohort 2, 15 patients with CLDN18.2-positive, HER2-negative gastric signet-ring cell carcinoma will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to sign a written Informed Consent Form (ICF) and to comply with protocol-specified visits and related procedures.

  2. Age was 18-75 years at the time of signing the ICF, and gender was unlimited.

  3. Has histopathologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the gastric/gastroesophageal junction (G/GEJ AC).

  4. No received systemic therapy. 5. Has histopathologically confirmed CLDN18.2-positive disease. 6. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.

Exclusion Criteria:

* 1. Has HER2-positive (defined as immunohistochemistry [IHC] 3+, or IHC 2+ and positive by in situ hybridization) disease.

  2. Is currently participating in another interventional clinical study, except when the subject is during survival follow-up of an interventional clinical study.

  3. Has a history of treatment with topoisomerase inhibitor-based antibody-drug conjugate(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  ORR is defined as the proportion of subjects in the analysis population who achieve confirmed objective response (CR or PR) as assessed by the IRRC per RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  Overall survival (OS) is defined as the time from enrollment to death from any cause.
Progression-free survival (PFS) | up to 2 years
  Progression-free survival (PFS) is defined as the time from enrollemnt to disease progression or death from any cause.
Disease control rate (DCR) | up to 2 years
  DCR is defined as the proportion of subjects in the analysis population who achieve disease control (CR, PR, or SD) as determined by the IRRC per RECIST v1.1 criteria.
Treatment-related adverse event (TRAE) | up to 2 years
  Safety evaluation, such as hematotoxicity, hepatotoxicity, and renal function lab test, done continuously during treatment and the level of serum creatinine will be evaluated by using CTCAE 5.0 during study.

CONTACTS AND LOCATIONS:
Overall Officials: Min Shi, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No